CLINICAL TRIAL: NCT04203485
Title: A Randomized, Open-Label, Controlled, Multicenter Phase III Study of Camrelizumab Combined With Apatinib Mesylate or Camrelizumab Alone Versus Platinum-based Chemotherapy for First-line Treatment in Subjects With PD-L1 Positive Relapsed or Advanced NSCLC
Brief Title: Camrelizumab Combined With Apatinib Mesylate or Camrelizumab Alone for First-line Treatment in Subjects With Programmed Death Ligand 1 (PD-L1) Positive Relapsed or Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-315
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: PD-L1 Positive Non-small Cell Lung Cancer
MeSH Terms: interventions — camrelizumab; apatinib; Pemetrexed; Injections; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Camrelizumab 200mg + Apatinib Mesylate 250mg (Experimental): Camrelizumab 200mg q2w ivgtt+ Apatinib Mesylate 250mg once daily po qd
  Interventions: Biological: Camrelizumab 200mg; Drug: Apatinib Mesylate 250mg
- Camrelizumab 200mg (Experimental): Camrelizumab 200mg q2w ivgtt
  Interventions: Biological: Camrelizumab 200mg
- Pemetrexed/Paclitaxel injection+ Carboplatin (Active Comparator): For non-squamous NSCLC: Pemetrexed disodium for injection + Carboplatin; For squamous NSCLC: Paclitaxel injection + Carboplatin
  Interventions: Drug: Pemetrexed disodium for injection; Drug: Paclitaxel injection; Drug: Carboplatin

INTERVENTIONS:
Biological: Camrelizumab 200mg — Camrelizumab 200mg q2w ivgtt
  Arms: Camrelizumab 200mg; Camrelizumab 200mg + Apatinib Mesylate 250mg
Drug: Apatinib Mesylate 250mg — Apatinib Mesylate 250mg po qd
  Arms: Camrelizumab 200mg + Apatinib Mesylate 250mg
Drug: Pemetrexed disodium for injection — Pemetrexed disodium for injection 500 mg/m2 q3w
  Arms: Pemetrexed/Paclitaxel injection+ Carboplatin
Drug: Paclitaxel injection — Paclitaxel injection 175 mg/m2 q3w
  Arms: Pemetrexed/Paclitaxel injection+ Carboplatin
Drug: Carboplatin — Carboplatin AUC 5 mg/mL/min q3w
  Arms: Pemetrexed/Paclitaxel injection+ Carboplatin

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of Camrelizumab (200mg,q2w) combined with Apatinib(250mg qd) in subjects with PD-L1 positive relapsed or advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have recurrent or advanced (Stage IIIB-IV) non-small cell lung cancer confirmed by histology or cytology.
2. No prior systemic treatment. Subjects who have received prior neo-adjuvant, adjuvant chemotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment free interval of at least 6 months from randomization since the last chemotherapy cycle.
3. Subjects should not have a previously detected activating Epidermal Growth Factor Receptor (EFGR) mutation or Anaplastic Lymphoma Kinase (ALK) fusion oncogene.
4. Subjects must have measurable disease by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST 1.1 criteria;
5. Freshly acquired samples or archived specimens within 6 months before randomization must be provided.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion Criteria:

1. Radiologically confirmed central squamous cell carcinoma.
2. Untreated central nervous system metastases (such as brain or meningeal metastases).
3. Pleural effusion, pericardial effusion, or ascites with clinical symptoms that need drainage
4. Past or present with idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, tissue pneumonia (eg bronchitis, occlusive vasculitis), drug-induced pneumonia, active pneumonia during CT screening, or objective evidence of severe impairment of lung function
5. Subjects with an active, known or suspected autoimmune disease. Patients with type I diabetes who are receiving a stable dose of insulin, hypothyroidism who only needs hormone replacement therapy, and skin diseases (such as eczema, vitiligo, or psoriasis) that do not require systemic treatment and do not have acute deterioration within 1 year before the screening period, are allowed.
6. Subjects with suspected active tuberculosis should be examined for chest X-rays, sputum, and ruled out by clinical signs and symptoms.
7. Uncontrolled Cardiac Symptoms or Diseases.
8. Subjects with high blood pressure who cannot be controlled well with antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg).
9. Arterial / venous thrombosis events, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism, occurred within the first 6 months of randomization.
10. Subjects who have previously received anti-PD-1 / PD-L1 monoclonal antibody, anti-cytotoxic T lymphocyte antigen-4 monoclonal antibody, or vascular endothelial growth factor receptor (VEGFR) small molecule inhibitor therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by Independent review committee (IRC) | up to 2 years
  Progression Free Survival, defined as the time from randomization to the first occurrence of disease progression as determined by IRC with use of Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) or death from any cause, whichever occurs first.
Overall survival | up to 2 years
  Overall survival is the time interval from the date of randomization to death due to any reason or lost of follow-up

SECONDARY OUTCOMES:
PFS assessed by investigator | up to 2 years
  Progression-Free-Survival
Objective Response Rate | At the time point of every 6 weeks，up to 2 years
  Objective Response Rate, determined using RECIST v1.1 criteria, defined as best overall response (complete or partial response) across all assessment time points
Disease Control Rate | At the time point of every 6 weeks，up to 2 years
  Disease Control Rate, determined using RECIST v1.1 criteria
Duration of Response | Up to 2 years
  Duration of Response, determined using RECIST v1.1 criteria
Time to Treatment Failure | Up to 2 years
  Time to Treatment Failure, defined as the time from randomization to treatment discontinuation.
Adverse Events and Serious Adverse Events | from the first drug administration to within 90 days for the last Camrelizumab dose
  Adverse Events and Serious Adverse Events

REFERENCES:
- [Derived] Zhou C, Wang Y, Zhao J, Chen G, Liu Z, Gu K, Huang M, He J, Chen J, Ma Z, Feng J, Shi J, Yu X, Cheng Y, Yao Y, Chen Y, Guo R, Lin X, Wang Z, Gao G, Wang Q, Li W, Yang X, Wu L, Zhang J, Ren S. Efficacy and Biomarker Analysis of Camrelizumab in Combination with Apatinib in Patients with Advanced Nonsquamous NSCLC Previously Treated with Chemotherapy. Clin Cancer Res. 2021 Mar 1;27(5):1296-1304. doi: 10.1158/1078-0432.CCR-20-3136. Epub 2020 Dec 15. PMID 33323401